CLINICAL TRIAL: NCT00501384
Title: Study for the Prevention of Ascites (SPA): Comparison of Fixed Doses of SR121463B Versus Placebo in the Reduction of Recurrence of Cirrhotic Ascites
Brief Title: Satavaptan Dose-Ranging Study in the Prevention of Ascites
Acronym: SPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI4522; LTS5635; LTS10209
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Ascites; Liver Cirrhosis
Keywords: cirrhotic ascites
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — satavaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: satavaptan (SR121463B)

SUMMARY:
The primary objective is to determine the optimal dose or range of doses of SR121463B for the reduction in recurrence of ascites, when used concomitantly with a standard dose regimen of spironolactone.

The secondary objective was to determine the tolerability of different fixed doses of SR121463B in cirrhotic ascites, over a 12-week treatment period.

This SPA study is followed by a single-blind, placebo-controlled, 40 weeks long-term safety extension (ExSPA). The first extension is followed by another long-term study (PASCCAL-1).

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of the liver confirmed by ultrasound, endoscopic examination or biochemical evidence
* Patients having undergone therapeutic paracentesis for the removal of ascites in the previous 24 hours with the removal of ≥4 L of fluid
* Patients having undergone at least 1 other therapeutic paracentesis in the previous 3 months

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2004-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Time to repeat therapeutic paracentesis | 12 weeks

SECONDARY OUTCOMES:
Increase in ascites judged by body weight and ascites volume | within 12 weeks
frequency of paracentesis | 12 weeks
quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Taipei, Taiwan

REFERENCES:
- [Derived] Wong F, Gines P, Watson H, Horsmans Y, Angeli P, Gow P, Minini P, Bernardi M. Effects of a selective vasopressin V2 receptor antagonist, satavaptan, on ascites recurrence after paracentesis in patients with cirrhosis. J Hepatol. 2010 Aug;53(2):283-90. doi: 10.1016/j.jhep.2010.02.036. Epub 2010 May 24. PMID 20541828
- See also: Related Info — http://www.sanofi-aventis.com